CLINICAL TRIAL: NCT02767219
Title: The Use of Bevacizumab as a Modulator of Wound Healing Following Trabeculectomy Surgery: A Single Centre Randomised Controlled Phase III Pilot Study
Brief Title: The Use of Bevacizumab as a Modulator of Wound Healing Following Trabeculectomy Surgery
Acronym: RAFTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MATR1001; 2013-000395-15 (EudraCT Number)
Record Dates: First submitted 2016-03-15; First posted 2016-05-10 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma
Keywords: Ophthalmology
MeSH Terms: conditions — Glaucoma | interventions — Bevacizumab; Fluorouracil; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone and 5-fluorouracil (Other): The control arm consists of current standard therapy of subconjunctival injections of dexamethasone 3.3mg/ml and pre filled syringes of 5-fluorouracil as required for 4 consecutive weeks after entry into the trial.
  Interventions: Drug: 5-fluorouracil; Drug: Dexamethasone
- Dexamethasone and Avastin (Active Comparator): Subconjunctival injections of dexamethasone 3.3mg/ml and pre filled syringes of bevacizumab will be given for 4 consecutive weeks from time of entry into trial
  Interventions: Drug: bevacizumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: bevacizumab — Patients will be randomised to study arms with a 1:1 ratio. Once randomised, Group 2 will receive a subconjunctival injection of bevacizumab and a subconjunctival injection of dexamethasone 3.3mg/ml. This will be given for 4 consecutive weeks from time of entry into trial.
  Other Names: Avastin
  Arms: Dexamethasone and Avastin
Drug: 5-fluorouracil — Patients will be randomised to study arms with a 1:1 ratio. Once randomised, Group 1 will receive a subconjunctival injection of 5-fluorouracil and a subconjunctival injection of dexamethasone 3.3mg/ml. This will be given as required for 4 consecutive weeks from time of entry into trial. This is current standard practice.
  Other Names: 5-FU
  Arms: Dexamethasone and 5-fluorouracil
Drug: Dexamethasone — Both intervention groups will be given a subconjunctival injection of dexamethasone at the time of injection of either bevacizumab or 5-fluorouracil

SUMMARY:
This is a phase III randomised controlled pilot study which aims to assess the effectiveness of the use of bevacizumab in patients who have undergone trabeculectomy surgery, which appear to be showing early signs of failure.

DETAILED DESCRIPTION:
Pharmacological enhancement of trabeculectomy using Mitomycin C (MMC) has significantly improved success rates. Despite this, some patients still mount aggressive scarring responses post-operatively and require additional subconjunctival injections of antifibrotic agents, such as 5-Fluorouracil (5-FU) to reduce scar formation and reduce the likelihood of surgical failure. There is concern that these agents are potentially toxic and may result in side effects such as keratopathy (loss of corneal epithelium) and are also painful for the patient. For those patients that are showing clinical evidence of potential scar formation, a more predictable and less toxic modulator of wound healing is desirable.

Vascular endothelial growth factor (VEGF) has been associated with angiogenesis in numerous pathological situations, including tumor growth, proliferative retinopathy, and rheumatoid arthritis. VEGF is also thought to play a pivotal role in ocular wound healing. It mediates the signal transduction cascade leading to tenon's fibroblast migration and proliferation and collagen gel contraction at the site of surgery, as well as angiogenesis. VEGF also causes persistent vascular permeability and vasodilation at the level of existing microvessels. Vessels with increased permeability are typically tortuous and dilated and this is the clinical appearance within the conjunctiva, suggestive of future excessive wound healing and scar formation following trabeculectomy. Early interventions such as subconjunctival injections of 5-Fluorouracil (5-FU) are therefore often considered when these clinical findings are apparent, in order to modify the course of wound healing.

The investigators propose a pilot study looking at the effect of serial injections of bevacizumab (an anti-VEGF agent) on modifying the wound healing response in patients showing early signs of future failure, compared to 5-Fluorouracil (5-FU). The purpose of the pilot is to also gather outcome data and information relating to safety and recruitment with a view to powering a definitive study addressing this issue.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years, inclusive
2. Patient must have undergone standard trabeculectomy augmented with Mitomycin C, within the past 4-6 weeks.
3. Patients who in the clinician's opinion are mounting an aggressive wound healing response and demonstrate objective increase in bleb vascularity (moderate or severe on MBGS). Bleb function still needs to be maintained in the clinicians opinion and flat, scarred blebs are not to be included.

Exclusion Criteria:

1. Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits.
2. Pregnant or nursing women.
3. A history of cardiovascular or cerebrovascular events in the previous 6 months, such as angina, arrhythmia, Transient Ischaemic Attack, strokes, myocardial infarction.
4. Uncontrolled hypertension defined as systolic blood pressure >160millimeters of mercury (mmHg) or diastolic blood pressure >90millimeters of mercury (mmHg)
5. Subject hypersensitive to bevacizumab, 5-Fluorouracil (5-FU), and Mitomycin-C (MMC) and its excipients
6. Failed trabeculectomy bleb
7. Persistent wound leak following trabeculectomy at the time of randomisation

   The following exclusions apply to the study eye only (i.e. they may be present for the non study eye
8. No light perception.
9. Aphakia
10. Previous, or planned, ocular surgery: vitreo-retinal, conjunctival surgery, etc considered likely to interfere with trabeculectomy outcome
11. Complicated cataract surgery
12. Cataract surgery less than 6 months in duration
13. Secondary glaucoma, other than Pigment Dispersion Syndrome (PDS) and Pseudoexfoliative (PXF)
14. Ocular trauma within the past 3 months
15. Active iris neovascularization or active proliferative retinopathy.
16. Severe posterior blepharitis.
17. Unwilling to discontinue contact lens use after surgery.
18. Current or recent (<3months) use of bevacizumab into the study eye.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Time taken to recruit 30 subjects (from start of study) | study start date to18 months
Proportion of patients who are eligible who agree to be randomized | study start date to 18 months
Proportion of patients who are lost to follow up or who withdraw from the study | Baseline to 36 months

SECONDARY OUTCOMES:
Intraocular pressure | Baseline to 18 months
Bleb morphology (as determined by Moorfields Bleb Grading system) | Baseline to 18 months
Number of additional postoperative interventions with 5-fluorouracil (5-FU) and subconjunctival dexamethasone, following the 4 week trial intervention period; bleb needling. | received between baseline and 18 months of follow up
Time to failure | Baseline to 18 months
Number of topical ocular hypotensive medications at 3 months and 18 months | 3 months and 18 months
The incidence of complications will be recorded: | Baseline to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Mathew, FRCOphthMBBS, Principal Investigator — Moorfields Eye Hospital NHS Trust; Jonathan Clarke, FRCOphthMBBS, Principal Investigator — Moorfields Eye Hospital NHS Trust; Keith Barton, FRCOphthMBBS, Principal Investigator — Moorfields Eye Hospital NHS Trust
Locations (1):
- Moorfields Eye Hospital, Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be disclosed publically, all the data will be anonymised and analysed in accordance with the Data Protection Act